CLINICAL TRIAL: NCT05635994
Title: Advanced Invasive Diagnosis (AID) Strategy for Patients With Chronic Coronary Syndromes Undergoing Coronary ANGIOgraphy (AID-ANGIO)
Brief Title: Advanced Invasive Diagnosis for Patients With Chronic Coronary Syndromes Undergoing Coronary ANGIOgraphy (AID-ANGIO)
Acronym: AID-ANGIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Responsible Party: Principal Investigator, Javier Escaned, Head of Interventional Cardiology, Hospital San Carlos, Madrid
Other Study IDs: 22/193-E
Record Dates: First submitted 2022-11-14; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Chronic Coronary Syndrome; Coronary Artery Disease; Microvascular Angina; Coronary Vasospasm; Myocardial Ischemia
Keywords: Chronic Coronary Syndrome; Microvascular Angina; Functional Coronary Angiography; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Microvascular Angina; Coronary Vasospasm; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: There is only one arm. Initially, a tentative diagnosis would be performed by the clinician, only taking into account patients's clinical information and angiography images. After applying AID strategy, a final diagnosis will be reached and compared with the tentative one.
  Interventions: Diagnostic Test: AID strategy

INTERVENTIONS:
Diagnostic Test: AID strategy — AID strategy encompasses a hierarchical algorithm intended to investigate both obstructive and non-obstructive causes of myocardial ischaemia. AID strategy starts with an ICA. Angiographically severe-grade stenosis (≥70%) can be safely considered flow-limiting without further physiological assessment. Conversely, by means of a pressure guidewire, intermediate-grade stenosis should be evaluated with FFR and/or NHPR in order to determine if they are physiologically significant. Those patients with non-obstructive CAD or normal epicardial coronary arteries should undergo functional coronary tests to investigate the presence of microcirculatory and vasomotor coronary disorders, which would account for non-obstructive causes of ischaemia.

SUMMARY:
AID-ANGIO is an observational, prospective, single arm, longitudinal study. Its objective is to investigate the diagnostic yield of the systematic use of a diagnostic strategy hierarchically addressing both obstructive and non-obstructive causes of myocardial ischaemia in an all-comers population of patients with chronic coronary syndromes (CCS) undergoing invasive coronary angiography (ICA). Angiographically severe-grade stenosis (≥70%) can be safely considered flow-limiting without further physiological assessment. Conversely, by means of a pressure guidewire, intermediate-grade stenosis would be evaluated with fractional flow reserve (FFR) and/or non-hyperaemic pressure ratios (NHPR) in order to determine if they are physiologically relevant. Those patients with non-obstructive CAD or normal epicardial coronary arteries would undergo functional coronary tests to investigate the presence of microcirculatory and vasomotor coronary disorders, which would account for non-obstructive causes of ischaemia. The main hypothesis of AID-ANGIO study states that, in patients with CCS referred to ICA, the application of a structured strategy -including ICA, physiological assessment of intermediate-grade stenosis and functional coronary tests- leads to a high diagnostic accuracy.

DETAILED DESCRIPTION:
AID-ANGIO is designed as an observational, prospective, single arm, longitudinal study, intended to assess the diagnostic yield of a hierarchical strategy which investigates both obstructive and non-obstructive causes of myocardial ischaemia in patients with CCS at the time of ICA. The diagnostic algorithm starts with an ICA. Angiographically severe-grade stenosis (≥70%) can be safely considered flow-limiting without further physiological assessment. Conversely, by means of a pressure guidewire, intermediate-grade stenosis should be evaluated with FFR and/or NHPR in order to determine if they are physiologically significant. Those patients with non-obstructive CAD or normal epicardial coronary arteries should undergo functional coronary tests to investigate the presence of microcirculatory and vasomotor coronary disorders, which would account for non-obstructive causes of ischaemia. The pressure guidewire to be used in the whole physiological evaluation (both epicardial and microvascular divisions) is the PressureWire X (Abbott) with a Coroventis Coroflow Cardiovascular System (Abbot) console.

After obtaining patients' informed consent, enrolment would encompass two steps. Firstly, a conventional ICA would be performed, according to standard practice. Then, obtained images would be displayed to patient's referring clinicians. They would be asked to identify epicardial stenosis affecting those vessels susceptible of revascularization, if they would be ≥ or <70%, and, in those <70%, if they would think they could be physiologically relevant. They would also be asked about the tentative therapeutic approach they would suggest, only taking into account patient's clinical information and ICA images. All this information would be collected in a written document to which the interventional team would be blinded. Subsequently, AID strategy would continue to be applied as previously described. Information gathered at the end of it would be written in a separated document by the interventional team. Next, referring physician and interventional team would together review the case, considering clinical information, ICA images and all findings from AID strategy application. Suitable cases for coronary artery bypass grafting (CABG), would also be discussed with a cardiovascular surgeon.

The AID-ANGIO study has a main hypothesis and two secondary hypotheses:

* Main hypothesis: In patients with CCS referred to ICA, the application of a structured AID strategy -including ICA, physiological assessment of intermediate-grade stenosis and functional coronary tests- leads to a high diagnostic accuracy.
* Secondary hypothesis (1): In patients with CCS referred to ICA, the application of a structured AID strategy leads to a significant change in their treatment.
* Secondary hypothesis (2): In patients with CCS referred to ICA, the application of a structured AID strategy increases the number of patients diagnosed with coronary microvascular dysfunction (CMD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with CCS, referred to ICA by their clinicians, suffering from angina and/or positive evidence of ischaemia in non-invasive tests and/or presence of CAD in computed tomography angiography.

Exclusion Criteria:

* Age <18 or >90 years old.
* Pregnancy.
* Severe left ventricle systolic dysfunction (LVEF ≤30%) or congestive heart failure.
* Any concomitant severe valve disease. Severely decreased renal function (glomerular filtration rate <30 mL/min/1.73 m2).
* Previous CABG.
* Presence of any anatomic features hampering intracoronary instrumentation with pressure guidewires.
* Contraindications to the administration of adenosine (asthma, 2nd or 3rd grade atrioventricular block without pacemaker, history of a non-ablationed accessory pathway-mediated tachycardia) or acetylcholine (asthma, 2nd or 3rd grade atrioventricular block without pacemaker, paroxysmal atrial fibrillation).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comer study population of patients with CCS referred to ICA.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a definite diagnosis of a cause of myocardial ischemia after ICA and an AID strategy. | From date of the first inclusion in the study until the date of last inclusion, assessed up to 48 months.
  To investigate the additional diagnostic value of an AID strategy over ICA alone in an all-comer population of patients with CCS.

SECONDARY OUTCOMES:
Number of patients in which the application of an AID strategy leads to a change from the initial treatment plan, only based in clinical information and ICA findings. | From date of the first inclusion in the study until the date of last inclusion, assessed up to 48 months.
  To investigate the influence of a structured AID strategy on the treatment plan in patients with CCS.
Number of patients with CMD, defined as low CFR or high IMR. | From date of the first inclusion in the study until the date of last inclusion, assessed up to 48 months.
  To study the prevalence of CMD in an all-comers population of patients with CCS referred to ICA.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Clinico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeronimo A, Paredes-Vazquez JG, Travieso A, Shabbir A, Jimenez-Quevedo P, Macaya-Ten F, Nombela-Franco L, Nunez-Gil IJ, Salinas P, Gomez-Polo JC, Garcia-Arribas D, Vilacosta I, Perez-Velasco JG, Garcia-Romo E, Garcia-Lledo A, Grande-Ingelmo JM, Fernandez-Rozas I, Alonso-Bello J, Curcio A, Fernandez-Ortiz AI, Villacastin JP, Mejia-Renteria H, Gonzalo N, Escaned J. Comprehensive diagnosis in chronic coronary syndromes combining angiography and intracoronary testing: the AID-ANGIO study. EuroIntervention. 2025 Jan 6;21(1):35-45. doi: 10.4244/EIJ-D-24-00499. PMID 39773829